CLINICAL TRIAL: NCT06654102
Title: A Controlled, Single Center Study to Evaluate the Cutaneous Effects of Deep Ultraviolet A (UVA) +/- High-Energy Visible (HEV) Blue Light Exposure
Brief Title: A Study to Evaluate the Cutaneous Effects of Deep Ultraviolet A +/- High-Energy Visible Blue Light Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CS2024SK100175
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Skin Pigmentation; Photobiology
Keywords: Skin Pigmentation; Photobiology
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Intervention Model Description: 4 test sites will be defined on the subjects' backs. Each test site will contain 7 subsites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regimen 1: Deep UVA (Experimental): Deep UVA, 380-400nm, will be used for subsites 2 to 7 of Test Sites 1 and 2.
  Interventions: Other: Deep UVA Irradiation
- Regimen 2: Deep UVA + HEV Blue Light (Experimental): Deep UVA + HEV Blue Light, 380-420 nm, will be used for subsites 2 to 7 of Test Sites 3 and 4
  Interventions: Other: Deep UVA+HEV Blue Light Irradiation
- Non-irradiated control (No Intervention): Subsite 1 in each test site (Test Sites 1-4) will be a non-irradiated control

INTERVENTIONS:
Other: Deep UVA Irradiation — A timed series of 6 UV doses will be administered to subsites 2 to 7 within Test Site 1 and 2 using an accurately calibrated solar simulator by varying the irradiation intensity for each subsite and keeping the duration of irradiation constant for all subsites. The duration of irradiation for each test site will be 30 minutes.
  Arms: Regimen 1: Deep UVA
Other: Deep UVA+HEV Blue Light Irradiation — A timed series of 6 UV doses will be administered to subsites 2 to 7 within Test Site 3 and 4 using an accurately calibrated solar simulator by varying the irradiation intensity for each subsite and keeping the duration of irradiation constant for all subsites. The duration of irradiation for each test site will be 30 minutes.
  Arms: Regimen 2: Deep UVA + HEV Blue Light

SUMMARY:
The objective of this study is to assess the level of pigmentation following an acute exposure of skin to light regimens representative of portions of the natural sunlight spectrum and that contain Deep UVA wavelengths with or without HEV Blue Light, as compared to non-irradiated control skin.

ELIGIBILITY:
Inclusion Criteria:

* Uniform skin color over the whole test area (the lower back) with minimal variation between test sites.
* At least 3 subjects per skin type, as defined by self-reported reaction to sun exposure and Chromameter measurements.
* Generally in good health.
* Able to read, write, speak, and understand English.
* Intends to complete the study and is willing and able to follow the subject responsibilities.

Exclusion Criteria:

* In another study without approval by the study site.
* Has known allergies or negative reactions to common topical skincare products or UV light.
* Has a history of abnormal responses to sunlight or UV radiation.
* Has used a tanning bed/lamp, has had extended sun exposure of the test area, or has participated in a UV exposure study within the past 4 weeks.
* Has a current illness/condition/situation, a medical history of a disease/condition, or a skin condition (e.g., psoriasis, rashes, eczema, seborrheic, severe excoriations, etc.) that could confuse the study results, interfere with participation, or increase health risk to the subject, as determined by the study investigator.
* Has shaved/waxed the test area within 2 weeks before Visit 1.
* Has used any products in the test area within 24 hours before Visit 1.
* Has sunburn, suntan, scars, tattoos, active dermal lesions, nevi, or other conditions in the test area that could confuse the study results or increase health risk to the subject, as determined by the study investigator.
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication.
* Is immunosuppressed (such as HIV-positive, transplant patients, undergoing chemotherapy or radiotherapy, etc.).
* Has been using a product or medication that the study investigator determines will increase health risk to the subject or confuse the study results
* Has a personal or family history of skin cancer.
* Skeletal protrusions and/or extreme areas of curvature in the test area.
* Is pregnant, nursing, or planning to become pregnant.
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Pigmentation level as determined by clinical evaluation | 15 mins and 18-22 hours Post-Irradiation
  The subsites of each test site will be graded for immediate or persistent pigmentation darkening (IPD/PPD) by a trained evaluator using a 0-2 grading scale, where 0 = no pigmentation darkening and 2 = moderate to intense pigmentation darkening.The mean values will be compared between each irradiated subsite and the non-irradiated subsite within the same test site and between each subsite in Regimen 1 compared to its corresponding subsite in Regimen 2.

SECONDARY OUTCOMES:
Pigmentation response as quantified by imaging | Baseline, 15 mins and 18-22 hours Post-Irradiation
  Images of each test site will be analyzed to quantify the level of pigmentation using L* and b* color space values, where an increase in pigmentation corresponds to a decrease in L* values and a potential decrease in b* values or increase in a* values. Change from baseline will be calculated. The mean values will be compared between each irradiated subsite and the non-irradiated subsite within the same test site and between each subsite in Regimen 1 compared to its corresponding subsite in Regimen 2.
Pigmentation response as quantified by Chromameter | Baseline, 15 mins and 18-22 hours Post-Irradiation
  A Chromameter will be used to quantify the level of pigmentation of subsites 1 and 7 using L* and b* color space values, where an increase in pigmentation corresponds to a decrease in L* values and a potential decrease in b* values or increase in a* values. Change from baseline will be calculated. The mean values will be compared between each irradiated subsite and the non-irradiated subsite within the same test site and between each subsite in Regimen 1 compared to its corresponding subsite in Regimen 2.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Union Research Center, a Division of SGS North America, Inc., Union City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No